CLINICAL TRIAL: NCT05288192
Title: Changes Noted After Suprachoroidal Triamcinolone Acetonide Injection.
Brief Title: Changes After Suprachoroidal Injection.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rc-3-22
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Retina; Change; Intraocular Pressure; Cataract; Macular Edema
MeSH Terms: conditions — Cataract; Macular Edema | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprachoroidal triamcinolone injection (Active Comparator): Eyes treated with suprachoroidal injection of triamcinolone acetonide.
  Interventions: Drug: Suprachoroidal triamcinolone acetonide (SCTA) injection
- Non-treated eyes (No Intervention): Eyes that are receiving no interventions during the study period.

INTERVENTIONS:
Drug: Suprachoroidal triamcinolone acetonide (SCTA) injection — Suprachoroidal injection of 4mg/0.1ml of triamcinolone acetonide.
  Other Names: SCTA injection
  Arms: Suprachoroidal triamcinolone injection

SUMMARY:
Changes after suprachoroidal injection are analyzed for statistical analysis.

DETAILED DESCRIPTION:
Changes after suprachoroidal injection of triamcinolone acetonide are noted in various retinal diseases treated by this technique to address its effects over six months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients prepared to suprachoroidal injection for various retinal diseases will be enrolled in the study.
* Bilateral retinal diseases that required interventions as diabetic macular edema, exudative retinal detachment, and serous chorioretinopathies.

Exclusion Criteria:

* Other retinal diseases that are not expected to improve after steroid injections as central retinal artery occlusion and age-related macular degenerations.
* Choroidal neovascularization that require anti-vascular endothelial growth factors.
* Patients refused to have steroid injections even after discussing the nature of their disease with them and the procedure to be done.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in visual acuity | Monthly after injection till six months of follow up
  Changes in best corrected visual acuity after injection
Changes in central foveal thickness | Monthly after injection till six months of follow up
  Changes in central macular thickness after injection

SECONDARY OUTCOMES:
Changes in intraocular pressure | Monthly after injection till six months of follow up
  Changes in intraocular pressure after injection
Changes in lens | Monthly after injection till six months of follow up
  Cataract progression after injection

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Tabl, MD, Principal Investigator — Benha University
Locations (1):
- Benha University, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: No